CLINICAL TRIAL: NCT05770284
Title: Effect of Exercise Based Regimen on Frailty in Children With Liver Disease -A Randomized Controlled Trial
Brief Title: Effect of Exercise Based Regimen on Frailty in Children With Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ILBS-Liver Disease-02
Record Dates: First submitted 2023-02-08; First posted 2023-03-15 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subject will receive 12 weeks of exercise with standard medical management (SMT) (Experimental): * Subjects will be given exercise protocol Pre-exercise safety assessment: Careful assessment as per exclusion criteria; especially Portal Hypertension, Cardiopulmonary status etc
  * Frequency: Aerobic and Resistance Exercises for total 50 minutes/day for 2-5 days per week (see protocol)
  * Aerobic exercises consist of Brisk walking
  * Resistance Exercises consist of movements targeting the major muscle groups with weight lifting
  * Intensity:
  Talk test: Short of breath but still can speak a full sentence Borg Scale: Keep between 5-6 out of 10.
  * Time duration of aerobic exercise decided by 6MWT, and resistance exercise by Hand grip strength
  * End point: 12 weeks
  * Stopping rule:
  * Interruption of Exercise for > 7 consecutive days due to non-compliance or clinical events.
  * Progression to exclusion criteria i.e. decompensation etc
  Both groups will be advised a calorie intake of 150cal/kg/day and protein intake of 3 gm/kg/day
  Interventions: Other: 12 weeks exercise; Other: Standard Medical Treatment
- standard medical management (SMT) (Active Comparator): standard medical management (SMT)
  Interventions: Other: Standard Medical Treatment

INTERVENTIONS:
Other: 12 weeks exercise — 12 weeks exercise
  Arms: Subject will receive 12 weeks of exercise with standard medical management (SMT)
Other: Standard Medical Treatment — Standard Medical Treatment

SUMMARY:
Frailty is now a well-known complication of liver disease and various studies, including pediatric literature studies, have recognized it as a poor prognostic factor in CLD as well as liver transplant settings. It is associated with poor quality of life, increased hospitalisation and mortality. Exercise for >12 weeks leads to improvements in aerobic power (peak VO2), aerobic endurance, muscle mass and strength, health related quality of life (HRQoL)(1). Although effect of Exercise on sarcopenia and frailty has been studied extensively in cirrhotic adults, there is paucity of such literature on the effect of exercise on frailty in children. Through this study, we aim to assess efficacy of exercise-based regimen on frailty in children with chronic liver disease after 12 weeks. Our secondary objective will be to compare outcome between the two groups(frail and non frail children with liver disease) and to compare change in frailty scores between the two groups. Other objectives will include assessment of the body composition analysis and the myokines and hepatokines signatures of children with liver disease (pre and post exercise intervention).

DETAILED DESCRIPTION:
Methodology Study population: Children with liver disease fulfilling the conditions as per inclusion and exclusion criteria

Baseline parameters that will be recorded:

* Clinical parameters:
* History and etiology of liver disease
* Symptomatology, Evidence of decompensation (jaundice, organomegaly, encephalopathy, ascites, infections, variceal bleed etc)
* PELD, MELD Na score, Lansky play performance score
* Baseline laboratory parameters: Complete blood count, LFT, KFT, PT-INR, ammonia etc
* Imaging parameters: liver and spleen size, portal vein size etc
* Anthropometric parameters:
* Weight for age
* Height for age
* BMI
* Triceps skin fold thickness
* Subscapular fold thickness
* Mid arm circumference

Calculation of frailty score:

Cut-off for frailty will be defined as frailty score >5 in children with liver disease.

Methodology for Frailty assessment:

Assessment of the 5 Fried Frailty Criteria would be performed at baseline in an ambulatory setting .The Fried Frailty assessment would be done in children with liver disease. The assessments will be typically performed by a combination of a doctor, dietician and physiotherapist.

Weakness-Grip strength would be measured using a handheld device, the Jamar Hand Dynamometer. The device would be squeezed 3 times by each hand, and the mean value of the recorded strength (in pounds) was taken as the final result and compared with standard values for age and sex. Slownessor endurance would be assessed by the 6-minute walk test (6-MWT). Children will use a standard hand wheel to capture the walked distance on a hard flat surface at their own pace. The covered distance expressed in meters (m) will be compared with standard values for sex and age. Shrinkage in children would be assessed by triceps skin fold thickness (TSF) measurements. TSF would be measured in triplicates by a dietician and the mean result was recorded in centimeters (cm) and compared with the Center for Disease Control age and sex normative values. Exhaustion-the Pediatric Quality of Life Inventory 4.0 Multidimensional Fatigue Scale, a validated pediatric questionnaire, would be used to assess fatigue. Diminished Physical activity-For children the age appropriate versions of the validated Modified Physical Activity Questionnaire (PAQ) (PAQ-A for children >13 years of age and PAQ-C for children< 13 yearof age will be used .

Along with routine investigations including Complete Blood counts, Liver function and Renal function test, PT-INR, serum Ammonia, the following investigations will also be done:

* Myokines (myostatin, decorin, irisin) and hepatokines (follistatin) levels in blood and urine at baseline and after 12 weeks of exercise therapy in study 2.
* Body composition analysis: Following parameters would be assessed: skeletal Muscle Mass; Body fat Mass; whole Body phase angle; segmental lean Analysis at baseline and after 12 weeks of exercise therapy in study 2.

Following enrolment and those fulfilling inclusion criteria, patient will then be allocated into exercise with SMT or SMT alone group as per block randomization method. Exercise with SMT or SMT alone will be given for a period of 12 weeks. Patient will be followed up for a period of 12 weeks. At the end of 12 weeks, frailty score will be recalculated .Body composition analysis,myokines and hepatokines will be repeated after 12 weeks.

Occurrence of clinical events including new onset ascites, AKI, hepatic encephalopathy, upper GI bleed and overall hospital stay as well as mortality over 12 weeks and 6 months will be noted in both groups during this period and treated as per standard of care. These events will be defined as follows-

1. Acute Kidney Injury

   As per KDIGO guidelines:
   * Increase in serum creatinine by more than 0.3mg/dl within 48 hours, OR
   * Urine output less than 0.5ml/kg/hour for more than 6 hours, OR
   * Increase in serum creatinine by more than 1.5 times the baseline presumed/known to have occurred within prior 7 days.
2. Hepatic encephalopathy: as per Modified West-Haven's criteria.
3. Grades of ascites Grade 1- ascites only detected by ultrasound Grade 2 -moderate ascites evident by distension of abdomen with shifting dullness Grade 3- gross/tense ascites with marked abdominal distension Study period: 2 years

Intervention (Study 2):

* Pre-exercise safety assessment: Careful assessment as per exclusion criteria; especially Portal Hypertension, Cardiopulmonary status etc
* Frequency: Aerobic and Resistance Exercises for total 50 minutes/day for 2-5 days per week (see protocol)
* Aerobic exercises consist of Brisk walking
* Resistance Exercises consist of movements targeting the major muscle groups with weight lifting
* Intensity:

Talk test: Short of breath but still can speak a full sentence Borg Scale: Keep between 5-6 out of 10.

• Time duration of aerobic exercise decided by 6MWT, and resistance exercise by Hand grip strength End point: 12 weeks

Stopping rule:

* Interruption of Exercise for > 7 consecutive days due to non-compliance or clinical events.
* Progression to exclusion criteria i.e. decompensation etc Both groups will be advised a calorie intake of 150cal/kg/day and protein intake of 3 gm/kg/day, and this will be ensured in regular follow-up as a standard care of practice developed by the department of Pediatric Hepatology.

Monitoring and assessment:

Patients will be followed up for a period of at least 3 months. Occurrence of clinical events including new onset ascites, AKI, hepatic encephalopathy, upper GI bleed, significant infections will be noted in both groups during this period and treated as per standard of care.

At the end of 12 weeks, frailty assessment will be repeated along with myokines and hepatokines, body composition analysis and anthropometric examination.

Adverse effects:

There are no expected adverse effects of exercise as seen in previous studies.

Stopping rule of study:

* Interruption of exercise for more than 7 consecutive days due to non-compliance or clinical events.
* Progression to exclusion criteria i.e decompensation
* Potential liver transplant within 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Children 9 - 18 years age with chronic liver disease & frailty score > 5.

Exclusion Criteria:

* Lansky play performance scale <50
* Unable to do exercise under supervision on at least 2 occasions
* Children on higher corticosteroid dose (>0.1mg/kg/day) in last 12 weeks
* Any degree of musculoskeletal involvement (myopathy/limb deformity/paraplegia)
* Children with any cardiac disease
* Children with neurological Wilson
* Uncontrolled portal hypertension (persistent high-risk varices) Recurrent variceal bleed ≥ 2
* Any degree of hemodynamic instability
* Current hepatic encephalopathy (any grade)
* Grade 3 ascites
* Hepatic hydrothorax
* Any degree of oxygen dependence
* Severe or Very severe Hepatopulmonary syndrome (room air PaO2 < 60 mm Hg).

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-11-02 (Actual); Study Completion 2024-11-02 (Actual)

PRIMARY OUTCOMES:
Prevalence of Frailty in children with liver disease. | 0 day
  Fraility assessment criteria will be based on 5 elements:
  1. weakness will be assessed by grip strength.
  2. slowness will be by 6 minutes walk test.
  3. shrinkage by triceps fold thickness.
  4. exhaustion by validated pediatric PedsQL 4.0 multidiamential fatigue scale.
  5. diminshed physical activity by modified PAQ
Improvement in Frailty after 12 weeks of exercise therapy in children with CLD and Frailty. | 12 weeks
  Improvement will be based on five fried fraility criteria with fraility score> 5

SECONDARY OUTCOMES:
Increase in skeletal muscle mass in Body composition analysis after 12 weeks of exercise regimen | 12 weeks
Decrease in the occurrence of Hepatic Encephalopathy based on modified West Haven criteria in the exercise regimen with SMT group versus SMT alone. | 3 months
Decrease in the occurrence of Upper Gastrointestinal bleed (presence or absence of GI bleed) in the exercise regimen with SMT group versus SMT alone. | 3 months
Decrease in the occurrence of significant events including Spontaneous Bacterial Peritonitis in the exercise regimen with SMT group versus SMT alone . | 3 months
Decrease in the occurrence of significant events including Acute Kidney Injury in the exercise regimen with SMT group versus SMT alone . | 3 months
Decrease in the occurrence of significant events including new onset or increase in ascites in the exercise regimen with SMT group versus SMT alone . | 3 months
Decrease in the occurrence of significant events including hospital stay in the exercise regimen with SMT group versus SMT alone . | 3 months
Decrease in the occurrence of significant events including mortality in the exercise regimen with SMT group versus SMT alone . | 3 months
Decrease in myostatin levels after 12 weeks of exercise regimen | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India